CLINICAL TRIAL: NCT01434823
Title: The Effects of 24-hour Intensivist Coverage in the Medical ICU
Brief Title: 24 Hour Intensivist Coverage in the Medical Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPenn 814063
Record Dates: First submitted 2011-08-30; First posted 2011-09-15 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2017-09

CONDITIONS: Critically Ill
Keywords: nocturnal staffing; intensivist staffing; intensivist coverage; ICU patient-centered outcomes; ICU resource utilization; patients admitted to the medical intensive care unit; Sleep Deprivation; Inattention; Work Hours
MeSH Terms: conditions — Critical Illness; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention - nocturnal coverage (Experimental): Nocturnal coverage from intensivists will be randomized by week. The weeks that have intensivists in the MICU during the 7pm to 7am shift are the intervention weeks.
  Interventions: Other: Nocturnal coverage
- Control - standard of care (No Intervention): The weeks that are not randomized, the intervention arm will retain the current standard of care in the HUP MICU: attending intensivist availability by phone (home call).

INTERVENTIONS:
Other: Nocturnal coverage — The investigators will randomize, by week, nocturnal coverage. During the intervention weeks, intensivists will be in the MICU from 7pm until 7am.
  For the Intensivist Sleep and Work sub-study:
  Measurements of Daytime Intensivist work hours, sleep, and attention will be measured with actigraphy, PVT, Sleep and Work Diaries, and Surveys. Results will be compared between periods with standard staffing to periods with overnight intensivist coverage.
  Arms: Intervention - nocturnal coverage

SUMMARY:
The Hospital of the University of Pennsylvania's Medical ICU (MICU) is implementing a model of 24-hour intensivist staffing in September 2011. Funds and resources are not available to cover the entire year, only certain weeks will be covered. The investigators propose a randomized clinical trial to study the comparative effectiveness of nocturnal intensivist staffing in the HUP MICU on patient outcomes. The investigators will be collecting and analyzing patient data of all patients admitted to the MICU from September 12, 2011, to September 11, 2012.

DETAILED DESCRIPTION:
Available evidence suggests that intensivist management of critically ill patients improves patient outcome, suggesting that greater intensivist coverage might be better still. However, the effects of 24-hour intensivist coverage in ICUs are unknown. In FY11, leadership of the Hospital of the University of Pennsylvania (HUP) decided to roll-out a program for partial night-coverage of the Medical Intensive Care Unit (MICU). In light of this natural experiment, the investigators propose to study the comparative effectiveness of nocturnal intensivist staffing in the HUP Medical Intensive Care Unit. To do so, the investigators propose a randomized clinical trial comparing the presence of a nocturnal intensivist (in-hospital call) to a traditional model of nocturnal coverage with an intensivist available by phone (home call) in the HUP MICU, with respect to patient-centered outcomes and resource utilization. The investigators will randomly assign seven consecutive days (Monday through Sunday) at a time to in-hospital or home call, in two-week blocks. The investigators will conduct primary analyses of all patients admitted during night hours and secondary analyses of various subgroups of patients admitted during night hours as well as all patients admitted during any time of day during the study period from September, 2011, to June, 2011.

A sub-study designed to measure sleep and work duration, sleepiness, and attention in Daytime Intensivists (faculty and fellows) during their medical ICU rotation will be conducted. The variables measured will be compared between periods with and without in-house nocturnal intensivist staffing. All fellows and faculty who rotate through the medical ICU during this study period, Jan 2012 to Dec 2012 will be approached for possible recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years and older, who are admitted to the HUP MICU during the 12-month study period will be included in the study.

Exclusion Criteria:

* No patients who meet these inclusion criteria will be excluded from this study.
* For patients admitted more than once to the MICU during the same hospitalization, we will include only their first admission to the MICU for all analyses.
* Subjects under 18 are very rarely seen at the HUP MICU because they are generally treated at the Children's Hospital of Philadelphia.
* In the rare event that a subject under the age of 18 receives care in the MICU his or her data will be excluded from this study.

For the Intensivist Sleep and Work sub-study looking at sleep, work hours, and attention of Daytime Intensivists during their MICU rotations:

* All University of Pennsylvania faculty members and fellows from the Division of Pulmonary, Allergy and Critical Care will be eligible for inclusion in the study if they rotate through the MICU during the study period (January, 2012 through December, 2012).

Exclusion Criteria:

* There are no exclusion criteria for this sub-study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1609 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Halpern, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bakhru RN, Basner M, Kerlin MP, Halpern SD, Hansen-Flaschen J, Rosen IM, Dinges DF, Schweickert WD. Sleep and Work in ICU Physicians During a Randomized Trial of Nighttime Intensivist Staffing. Crit Care Med. 2019 Jul;47(7):894-902. doi: 10.1097/CCM.0000000000003773. PMID 30985450
- [Derived] Kerlin MP, Small DS, Cooney E, Fuchs BD, Bellini LM, Mikkelsen ME, Schweickert WD, Bakhru RN, Gabler NB, Harhay MO, Hansen-Flaschen J, Halpern SD. A randomized trial of nighttime physician staffing in an intensive care unit. N Engl J Med. 2013 Jun 6;368(23):2201-9. doi: 10.1056/NEJMoa1302854. Epub 2013 May 20. PMID 23688301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled all patients admitted to the medical ICU (MICU) service at the Hospital of the University of Pennsylvania for one year from September 12, 2011, to September 11, 2012. In-hospital follow-up was conducted for an additional 90 days.
Pre-assignment Details: Exclusions included patients who were readmitted to the ICU within the same hospitalization (we included their first ICU admission), patients who were admitted during the holiday block (no nighttime coverage), and patients who had ICU stays so brief they were either were not exposed to nighttime hours or ineligible for APACHE score calculation.
Groups:
- Intervention - Nocturnal Coverage: Nocturnal coverage from intensivists will be randomized by week. The weeks that have intensivists in the MICU during the 7pm to 7am shift are the intervention weeks.
  Randomization was blocked such that 1 week of a 2-week attending block of service was randomized to nocturnal coverage. We also calculated the proportion of "covered nights" for each patient's ICU stay in secondary analyses.
- Control - Standard of Care: The weeks that are not randomized, the intervention arm will retain the current standard of care in the HUP MICU: attending intensivist availability by phone (home call).
  Randomization was blocked such that 1 week of a 2-week attending block of service was randomized to nocturnal coverage. We also calculated the proportion of "covered nights" for each patient's ICU stay.
Period: Overall Study
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Started | 824 | 785
Completed | 820 | 778
Not Completed | 4 | 7
Not completed — Incomplete data in medical record | 4 | 7

BASELINE CHARACTERISTICS:
Population: 824 patients were randomized to the intervention group, 4 of which have been excluded from analyses to due incomplete data (n=820), 785 were randomized to the control group, 7 of which have been excluded from analyses due to incomplete data (n=778).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care | Total
Number analyzed (Participants) | 820 | 778 | 1598
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (17) | 59 (16) | 58 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 366 | 356 | 722
  Male | 454 | 422 | 876
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 11 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 328 | 315 | 643
  White | 417 | 387 | 804
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 70 | 65 | 135
Region of Enrollment [Number; unit: participants]
  United States | 820 | 778 | 1598

OUTCOME MEASURES:

1. Primary Outcome: MICU Length of Stay
Description: Time from ICU admission to discharge
Time Frame: From time of admission in the MICU until time of discharge from the MICU - assessed up to 12 months
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Number analyzed (Participants) | 820 | 778
hours | 52.8 [29.3 to 116.1] | 52.6 [28.2 to 110.5]

2. Secondary Outcome: MICU Mortality
Description: Mortality will be assessed during each patient's stay in the MICU from admission to discharge
Time Frame: From time of admission to MICU until discharge from MICU - assessed up to 12 months
Measure: Number; unit: participants
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Number analyzed (Participants) | 820 | 778
participants | 154 | 139

3. Secondary Outcome: In-hospital Mortality
Description: Mortality will be assessed during each patient's stay in the hospital.
Time Frame: From time of admission to MICU to hospital discharge - assessed up to 12 months
Measure: Number; unit: participants
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Number analyzed (Participants) | 820 | 778
participants | 203 | 177

4. Secondary Outcome: Re-admission to the MICU Within 48 Hours
Description: The investigators will measure, in hours, the time spent from discharge from the MICU until a patient is re-admitted to the MICU during the same hospital stay.
Time Frame: From time of discharge from MICU, to re-admission to the MICU - assessed up to 12 months
Measure: Number; unit: participants
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Number analyzed (Participants) | 820 | 778
participants | 32 | 21

5. Secondary Outcome: Discharge Home From Hospital
Description: Patients who were discharged from the hospital to their homes
Time Frame: Assessed up to 12 months
Measure: Number; unit: participants
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Number analyzed (Participants) | 820 | 778
participants | 317 | 314

6. Secondary Outcome: Daytime Intensivist Daily Sleep Duration
Description: This will be the primary outcome of the Intensivist Sleep and Work sub-study.
Time Frame: Daily
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Intervention - Nocturnal Coverage: Nocturnal coverage from intensivists will be randomized by week. The weeks that have intensivists in the MICU during the 7pm to 7am shift are the intervention weeks.
  Nocturnal coverage: The investigators will randomize, by week, nocturnal coverage. During the intervention weeks, intensivists will be in the MICU from 7pm until 7am.
  For the Intensivist Sleep and Work sub-study:
  Measurements of Daytime Intensivist work hours, sleep, and attention will be measured with actigraphy, PVT, Sleep and Work Diaries, and Surveys. Results will be compared between periods with standard staffing to periods with overnight intensivist coverage.
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Number analyzed (Participants) | 20 | 20
hours | 6.69 (0.13) | 6.37 (0.16)

ADVERSE EVENTS:
Arm/Group | Intervention - Nocturnal Coverage | Control - Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/820 | 0/778
Other Adverse Events (participants affected / at risk) | 0/820 | 0/778

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No